CLINICAL TRIAL: NCT06833606
Title: Diagnosis and Outcomes of Placental Accretism
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PLC_AC
Record Dates: First submitted 2024-12-03; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Placenta Accreta
Keywords: diagnosis
MeSH Terms: conditions — Placenta Accreta; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the diagnostic ability of the main criteria currently adopted for the diagnosis of placenta accreta and to define the maternal outcomes in terms of complications of the different management strategies currently adoptable when placental accretism is suspected.

DETAILED DESCRIPTION:
Currently, the management of cases of placental accretism/percretism is not standardized. This study could help in assessing maternal and fetal outcomes related to the different therapeutic strategies applied in the clinical cases under study so that their management can be standardized in the near future.

This is a retrospective and prospective, national multicenter study. Patients will be treated according to clinical practice.

The main instrumental findings of cases of suspected accretism will be collected and analyzed, and the progression of pregnancy and postpartum (by means of laboratory and instrumental tests) will be evaluated in order to define the outcomes of conservative management (cesarean section with placenta in situ) versus more radical management (cesarean section and concomitant hysterectomy).

In particular, clinical trends (by means of assessment of vital parameters, laboratory tests, ultrasound images or instrumental examinations) in pregnancy, in the immediate postoperative period and during subsequent outpatient follow-up visits will be analyzed.

In general, in the absence of complications, visits will be performed twice a week during pre-partum. Postpartum follow-up is not standardized, as it will depend strictly on the procedure performed and the occurrence or absence of complications. There are no questionnaires and/or rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 44 years
* Pregnant women with suspected placental accretism
* Acquisition of informed consent form

Exclusion Criteria:

None

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with suspected placental accretism/percretism followed at the Outpatient Clinics of the Division of Obstetrics and Prenatal Age Medicine at IRCCS-AOUBO Policlinico di Sant'Orsola and participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of correspondence between prenatal diagnosis and intra-operative finding of placental accretism | Up to 1 month post-partum
  disappearance of the hypoecogenaretroplacental stria, lacunae placental vasculature, hypervascularization of the utero-vesical interface, interruption/irregularity of the bladder will be assessed by ultrasound

SECONDARY OUTCOMES:
Frequency of maternal complications (Surgical site infection) | Up to 1 month post-partum
  Post-operative haemorrhage and haemotransfusion, infection of the surgical site will be assessed by blood count with leucocyte formula, coagulation tests (thrombin time, thromboplastin time and fibrinogen), PCR (C-reactive protein), blood cultures

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Pilu, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (7):
- Italy (7):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Ospedale "M. Bufalini", Cesena, Forlì-Cesena
  - Ospedale "Morgagni-Pierantoni", Forlì, Forlì-Cesena
  - AOU Policlinico di Modena, Modena, Modena
  - Azienda Ospedaliero - Universitaria di Parma, Parma, Parma
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Reggio Emilia
  - Ospedale "Infermi" di Rimini, Rimini, Rimini